CLINICAL TRIAL: NCT06446908
Title: Acceptability and Feasibility of a New Approach to Engage Patients With Steatotic Liver Disease in Physical Activity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Montfort (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-A06PHYSACTIV
Record Dates: First submitted 2024-05-27; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Liver Steatosis; MASH; MASLD
Keywords: Physical activity; coaching; telehealth; liver
MeSH Terms: conditions — Fatty Liver; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coaching Intervention (Experimental): This study is an open-label, mono-centred, single-case experimental design with multiple base levels. The study will comprise 3 phases, alternating periods of observation (A) and 1 period of counselling (B) with an A1-B-A2 design.
  PA will be assessed continuously using an accelerometer for 7 to 14 days per (A) phase. During phase (B), participants will receive the intervention, i.e. 6 x 45-minute, real-time, face-to-face, virtual sessions with a PA counsellor.
  Interventions: Behavioral: Telehealth coaching for liver disease

INTERVENTIONS:
Behavioral: Telehealth coaching for liver disease — This study is an open-label, mono-centred, single-case experimental design with multiple base levels. The study will comprise 3 phases, alternating periods of observation (A) and 1 period of counselling (B) with an A1-B-A2 design.
  PA will be assessed continuously using an accelerometer for 7 to 14 days per (A) phase. During phase (B), participants will receive the intervention, i.e. 6 x 45-minute, real-time, face-to-face, virtual sessions with a PA counsellor.

SUMMARY:
Steatosis is the building of fat in the liver. Steatotic liver disease (SLD) regroups MASLD (metabolic dysfunction-associated steatotic liver disease) and MASH (metabolic dysfunction-associated steatohepatitis) i.e. MASLD with inflammation. An estimated 30% of the population worldwide has MASLD and 5% of Canadians have MASH. MASH is a leading cause of liver transplantation in Canada. There is no cure for SLD, and the treatment relies on diet, weight loss, and physical activity (PA).

Is a counselling intervention to help patients progressively engage in more PA a feasible and acceptable approach? Objectives. This proposal has three primary objectives: 1) To assess the feasibility of our PA counselling intervention (to be delivered online) with SLD patients; 2) To evaluate the acceptability of our intervention; 3) To evaluate the feasibility of the study methods/procedures.

Methodology. This study is an open-label, mono-centred, single-case experimental design with multiple base levels. The study will comprise 3 phases, alternating periods of observation (A) and 1 period of counselling (B) with an A1-B-A2 design.

PA will be assessed continuously using an accelerometer for 7 to 14 days per (A) phase. During phase (B), participants will receive the intervention, i.e. 6 x 45-minute, real-time, face-to-face, virtual sessions with a PA counsellor.

Based on past studies, our sample size will be 12 participants. They will be recruited through the hepatology clinic at Hôpital Montfort.

The primary outcomes of the project are to evaluate the feasibility and acceptability of the trial and intervention. The secondary outcomes are Daily PA time and biological/imaging data evolution

DETAILED DESCRIPTION:
Background and rationale: This pilot trial aims to evaluate the feasibility and acceptability of a counselling intervention on physical activity in patients with liver steatosis (primary aim) and changes in molecular outcomes (exploratory aim).

Liver steatosis is the build-up of fat in the form of lipid droplets inside hepatocytes (liver cells). Although it is a form of energy storage, it is considered pathological when more than 5% of hepatocytes demonstrate fat infiltration on a liver biopsy or imaging (ultrasound, magnetic resonance, or computed tomography). Until recently, liver steatosis was described as two entities with a clinicopathological continuum: non-alcoholic fatty liver disease (NAFLD) and non-alcoholic steatohepatitis (NASH) i.e. NAFLD with inflammation. NAFLD/NASH is strongly associated with features of the metabolic syndrome: type 2 diabetes mellitus (DM), hyperlipidemia, and obesity. Insulin resistance is considered one of the first steps to developing fatty liver infiltration. Indeed, 70% to 80% of patients with diabetes have NASH. A recent change in nomenclature now accounts for the link with cardiometabolic criteria. NAFLD is now MASLD (metabolic dysfunction-associated steatotic liver disease) i.e. steatosis and at least 1 cardiometabolic factor and NASH is MASH (metabolic dysfunction-associated steatohepatitis) i.e. MASLD with inflammation, regrouped as steatotic liver disease (SLD).

SLD is a silent disease: patients have no symptoms, are not routinely screened for the disease, and SLD is often revealed through complications of cirrhosis, at a late stage for intervention. Inflammation is confirmed when liver function tests alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are elevated. It is recommended to assess the level of associated fibrosis through non-invasive tests such as elastography that evaluates liver stiffness that increases with fibrosis, or algorithms such as Fibrosis-4 (FIB-4) that combines age, ALT, AST, and platelets count to identify fibrosis in patients over 35 years old. The SLD burden is expected to increase. An estimated 30% of the population worldwide has MASLD and 5% of Canadians have MASH (2). A Canadian study concluded that the number of people with post-MASH decompensated cirrhosis will double by 2030 and cases of liver cancer will increase by 80 % (2). MASH is a leading cause of liver transplantation in Canada (2). Despite extensive research with currently over 1350 active clinical trials (clinicaltrials.gov, accessed 19/09/2023), there is no cure for SLD, and the treatment relies on diet, weight loss, and physical activity (PA). The current North American guidelines state that patients with NAFLD should be strongly encouraged to engage in PA to the extent possible.

The effects of PA on SLD have been studied extensively. A systematic review (3) showed personalized PA improved the quality of life for cirrhotic patients without significant side effects and may reduce the 90-day readmission rates for transplant patients at the end of the program. Henri et al. showed US NAFLD adults who engaged in vigorous PA have a lower risk of death from cancer and all causes than NAFLD adults who do not engage in any PA; benefits persisted for low PA and any PA versus no PA (4). Similarly, a US study showed PA is inversely associated with NALFD and associated with better survival for NALFD patients (5). PA is also successful in preventing DM, which is now included in the MASH definition (6). Moreover, meta-analyses have concluded that PA contributes to decreasing levels of various biological markers of SLD (7), (8) and inflammatory markers (9), thus reducing intra-hepatic fat (10), (11), (12), (13). PA is thus efficacious in reducing inflammation and fibrosis in patients with SLD. However, key knowledge gaps remain including (1) scarce data on the impact of sustained PA in MASH patients, especially post-participation in studies, (2) lack of consistency in terms of eligibility criteria that are often too narrow and exclude patients seen in practice, (3) heterogeneous PA parameters (e.g., dosage, type, duration), and (4) variability of biological data collected. It is thus difficult to precisely define through meta-analyses and/or systematic reviews the optimal program to help support PA or its duration. Another critical gap is what is the influence of interventions that aim to have patients initiate and maintain PA on their own. This is important because in reality, it is not possible (or sustainable) to offer patients supervised PA sessions in the amount that is commensurate with current PA guidelines, considering patients have their own barriers to PA and the lack of support to help them initiate and maintain PA in everyday life. Indeed, from discussions with patients during clinical evaluation with Dr. Fresne, some barriers are lack of time, insufficient knowledge, fear of injury, and lack of financial resources. In the literature, perceived lack of resources and education, physical discomfort or limitations or pain, lack of space, and time constraints have been identified as barriers for PA (13),(14), (15).

We believe individualized support and guidance to help patients progressively engage in more PA is a better results-oriented sustainable approach than delivering supervised PA training sessions and propose a personalized counselling intervention to engage patients with SLD in PA.

Additionally, whether having patients initiate and maintain PA in everyday life by providing them with support can contribute to reducing inflammation and/or fibrosis in the liver remains to be described. It is known that sarcopenia (loss of skeletal muscle mass and strength) is associated with cirrhosis/liver fibrosis and DM, suggesting communication between the liver and muscles. During PA, the muscle secretes small peptides called myokines that act on the skeletal muscle, but also on distant organs, to improve their function, including decreasing inflammation and liver lipid content, such as interleukin 6 (IL-6), IL-15, irisin (16). PA also modifies the secretion of hepatokines, peptides secreted by hepatocytes. It is therefore possible that levels of these proteins will be modified in our population if they can initiate and maintain PA during their participation in PA counselling compared to their baseline PA level. These proteins could therefore serve as biomarkers to determine the efficacy of the PA counselling in improving SLD and reducing inflammation.

Significance and Innovation:

Engaging SLD patients in PA is crucial and a matter of public health. The number of SLD patients will increase in the next 10 years and there is currently no medication to treat the condition nor prevent the evolution towards cirrhosis with the associated risk of liver transplant and cancer. PA has proven its efficacy in SLD. However, physicians may not know how to help their patients to practice PA as a treatment and SLD patients face barriers to PA that need better characterization. We believe our innovative PA intervention using personalized counselling could help patients to overcome their barriers to PA. To our knowledge, this would be the first study that would provide patients keys to successfully engage in PA and empower SLD patients with PA through counselling. We believe participants in our study will be more likely to maintain long-term PA and the project will help us understand the barriers and facilitators to PA behavior change faced by SLD patients. If this feasibility project proves successful, we will develop a larger trial to assess the long-term engagement of SLD patients in PA and study the effects of PA on the interaction between liver, fat, and muscle in SLD patients.

Population and recruitment: Based on past SCED studies, our sample size will be 12 participants. They will be recruited through the hepatology clinic at Hôpital Montfort.

Intervention: The intervention is informed by the Telehealth Bariatric Behavioral Intervention (TELE-BariACTIV) study led by Drs Baillot and Brunet (18). The TELE-BariACTIV has been developed to increase PA for patients awaiting bariatric surgery. It is based on the principles of the BariACTIV trials (19),(20) that demonstrated a 6-week period of personalized face-to-face counselling before surgery centered on behavioral strategies such as goal-setting and self-monitoring significantly increased pre-surgery moderate-to-vigourous PA. TELE-BariACTIV was designed to reinforce theory-based content and participant's perspective, and include telehealth to increase reach. It was successfully tested (article in preparation) using a SCED. The purpose of the intervention is to increase autonomy, motivation, and self-confidence so participants can autonomously engage in PA. The content of the TELE-BariACTIV counselling is meant to be adapted to reflect participants' conditions, and we will do so by working with a patient-partner. The intervention aims to increase motivation (via satisfaction of basic psychological needs) and self-efficacy, critical determinants of PA behavior change.

Data collection: We will collect sociodemographic data such as age, sex, gender, language, level of education, profession, and income. PA will be measured daily throughout the trial via an accelerometer (7-14 days in each (A) phase) mailed to the participants. They will be instructed to wear the accelerometer continuously, except during water-based activities, and to maintain a log of wear times with waking and bed times. Accelerometer data will be extracted and downloaded (10-second epochs) using the appropriate software and will be cleaned in accordance with the logbooks provided by the participants.

Qualitative data: We will collect data on (1) participants' opinions of the trial (assessments, timing, etc.) and intervention via with a semi-structured interview at the end of their participation, (2) onacceptability with a 7-item questionnaire developed and validated by the research team, and (3) on PA counsellor notes for each intervention session, for examples, duration, topics discussed, accomplishment of session objectives, participants' reactions to the content, next steps with the participants, and reflections as a PA counsellor (e.g., problems arising during the sessions, overall experience delivering the session, suggestion for intervention or personal improvements, and session deviations).

Quantitative data: We will collect/measure pre and post intervention data for : liver function tests (ALT, AST, Gamma Glutamyl Transferase, Alkaline Phosphatase, bilirubin, albumin), total/High Density Lipoprotein/Low Density Lipoprotein cholesterol levels, triglycerides levels, fasting glucose and insulin, HbA1c, fasting free fatty acids, Body Mass Index, waist circumference, IL-6, TNF-α, CReactive Protein, and leptin, and calculate composite scores such as FIB-4. We will also evaluate liver fibrosis with a liver elastography before screening and at the end of participation. Myokines and hepatokines will be measured using available kits.

Data analysis:

Quantitative data: Descriptive statistics will be computed for baseline sociodemographic, clinical, biological, feasibility, and acceptability data derived from the numerical responses and close-ended questions. All statistical analyses will be carried out using R and the appropriate packages. A Tau-U test for each participant and for the group will be performed to compare daily PA based on accelerometer data between phases A1 and B, as well as A1 and A2. Individual effect sizes will be aggregated in a meta-analysis to obtain a group-based effect size. A sensitivity analysis will also be performed with a randomization test.

Qualitative data: The content of the interviews and the PA counselors' notes completed after the sessions will be analyzed by two team members using content analysis after verbatim transcription, using the NVivo software.

Based on data from the TELE-bariACTIV study, our project will be deemed successful if the refusal rate is ≤25%, the retention rate after phase B (PA intervention) is ≥75%, the intervention attendance rate is ≥75%, and the intervention attrition rate ≤25%. The main objectives of our project are feasibility and acceptability: at this point, the evolution or lack of evolution of biological or imaging markers before and after participation will not be considered for the success of the project. It will, however, help define which markers should be used for a large-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age,
* confirmed MASLD or MASH without cirrhosis
* access to a computer with an internet connection

Exclusion Criteria:

* liver disease from another cause,
* the existence of cirrhosis on imaging or clinically,
* weekly alcohol consumption over 50g,
* having a contraindication to PA without medical clearance (the Get Active questionnaire from the Canadian Society for Exercise Physiology is used to determine if medical clearance is needed),
* being already enrolled in a supervised exercise intervention or PA behaviour change intervention or currently meeting PA guidelines of 150 mins/week
* the need for a wheelchair, cane, walker, or other support(s) to move

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
attendance rate of participants | 1 year
  to evaluate the feasibility of the intervention
number of participants who completed the intervention | 1 year
  to evaluate the feasibility of the intervention
refusal rates | 1 year
  to evaluate the feasibility of the trial
recruitment rates | 1 year
  to evaluate the feasibility of the trial
attrition rates | 1 year
  to evaluate the feasibility of the trial
semi-structured interviews at the end of participation | 18 months
  to evaluate the acceptability of the intervention
7-item questionnaire developed for the TELE-BariACTIV study with statements in the future tense for before phase B or past tense for after phase B | 18 months
  to assess retrospective and prospective acceptability

SECONDARY OUTCOMES:
Measurement of daily PA time using a accelerometer during phases A | 18 months
  to evaluate the changes in daily PA before and after the coaching intervention
Measurement of liver function tests (ALT, AST, Gamma Glutamyl Transferase, Alkaline Phosphatase, bilirubin, albumin) | 18 months
  to evaluate the changes in biological variables before and after the coaching intervention
Measurement of lipids : fasting free fatty acids, total/High Density Lipoprotein/Low Density Lipoprotein cholesterol levels, triglycerides levels | 18 months
  to evaluate the changes in biological variables before and after the coaching intervention
Measurement of glucose levels: fasting glucose and insulin, HbA1clevels, triglycerides levels | 18 months
  to evaluate the changes in biological variables before and after the coaching intervention
Measurement of weight | 18 months
  to evaluate the changes in BMI before and after the coaching intervention
Measurement of height | 18 months
  to evaluate the changes in BMI before and after the coaching intervention
Measurement of inflammation markers :IL-6, TNF-α, CReactive Protein, and leptin | 18 months
  to evaluate the changes inflammation markers before and after the coaching intervention
Measurement of elastography | 18 months
  to evaluate the changes liver fibrosis before and after the coaching intervention

CONTACTS AND LOCATIONS:
Overall Officials: Celine Fresne, MD, Principal Investigator — H[opital Montfort

IPD SHARING:
Plan to Share IPD: No